CLINICAL TRIAL: NCT05689775
Title: Reconstruction After Abdominoperineal Resection With Robot-assisted Harvest of VRAM Flap
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Frich, Consultant, Oslo University Hospital
Other Study IDs: 387180
Record Dates: First submitted 2022-11-23; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Perineum; Wound; Postoperative Complications; Rectal Neoplasms; Rectus Abdominis Hernia; Prospective Studies; Wound Heal; Sexual Health
Keywords: Rectus abdominis muscle flap; Reconstruction; Perineum
MeSH Terms: conditions — Wounds and Injuries; Postoperative Complications; Rectal Neoplasms | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients over 18 years of age operated for locally advanced anal or rectal cancer with robot-assisted abdomino-perinal resection and robot-assisted reconstruction of pelvic floor and/or vagina with vertical rectus abdomínis muscle flap.
  Interventions: Procedure: Reconstruction with robot-assisted rectus abdominis muscle flap

INTERVENTIONS:
Procedure: Reconstruction with robot-assisted rectus abdominis muscle flap — Reconstruction of perineum and/or vagina with robot-assisted rectus abdominis muscle flap.

SUMMARY:
Non-randomized study of robot-assisted perineal reconstruction with rectus abdominis muscle flap in patients operated with abdominoperineal resection for irradiated locally advanced rectal or anal cancer. Operative time, complications, wound healing, pre- and postoperatively abdominal wall strength and patient related outcomes including sexual health will be registered.

DETAILED DESCRIPTION:
Inclusion criteria:

Patients > 18 years of age operated with robotic-assisted abdominoperineal resection for irradiated locally advanced rectal or anal cancer where robotic-assisted perineal and/or vaginal reconstruction has been performed with a rectus abdominis muscle flap.

Methods Up to 40 patients operated with robotic-assisted abdominoperineal resection with Da Vinci Xi surgical system (Intuitive Surgical, Sunnyvale, California, USA) and robotic-assisted reconstruction with a pedicled rectus muscle will be included in this prospective, non-randomized study.

In addition to the standardized post-operative care for patients with locally advanced rectal or anal cancer as specified by national guidelines, patients will be offered study-specific follow-up visits at 1, 6 and 12 months.

Complications are recorded by the accordion severity grading system of surgical complications. Patient related outcomes measures will be registered by using European organization for research and treatment of cancer Quality of life questionnaire Core 30 (EORTC QLQ-C30). Sexual health will be registered by a subset of questions from European organization for research and treatment of cancer Quality of life questionnaire Sexual health (EORTC QLQ-SH22).

Primary endpoint:

- perineal wound healing at 3 months

Secondary endpoints:

* early (< 30 days) and late (> 30 days) complications
* quality of life preoperatively and at 3- and 12 months postoperatively
* sexual function preoperatively and at 3- and 12 months postoperatively
* clinical evaluation of abdominal wall strength preoperatively, at 3- and 12 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* patients with rectal or anal cancer
* scheduled for robot-assisted abdominoperineal resection
* reconstruction of pelvic floor and/or vagina with rectus abdominis muscle flap

Exclusion Criteria:

* patients not eligible for robot-assisted procedure
* rectus abdominis muscle not available for harvest
* the expected wound defect is not suitable for reconstruction with rectus abdominis muscle flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal or anal cancer who are scheduled for robot-assisted abdominoperineal resection who need reconstruction of pelvic floor and/or vagina with rectus abdomens muscle flap.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perineal wound healing | 3 months
  Perineal wound healing at 3 months.
  Perineal wound has completely healed at clinical control 3 months postoperatively without need for further follow-up of the perineal wound.
  Any perineal complications are noted.
  * superficial wound infection
  * deep wound infection
  * minor wound dehiscence
  * major wound dehiscence
  * partial flap loss
  * total flap loss
  * perineal hernia
  * enterocutaneous fistula
  * stricture in neovagina
  * perineal wound dehiscence not related to flap
  * other complications

SECONDARY OUTCOMES:
Early postoperative complications | Within 30 days postoperatively
  Early postoperative complications at 30 days.
  A. Abdominal/donor-site complications
  * superficial wound infection
  * deep wound infection
  * minor wound dehiscence
  * major wound dehiscence
  * abdominal hernia
  * other complications
  B. Perineal complications
  * superficial wound infection
  * deep wound infection
  * minor wound dehiscence
  * major wound dehiscence
  * partial flap loss
  * total flap loss
  * perineal hernia
  * enterocutaneous fistula
  * stricture in neovagina
  * perineal wound dehiscence not related to flap
  * other complications
  C. Other complications
  * incisional hernia
  * parastomal hernia
  * reoperation
  * other complications
  Complications are classified as mild, moderate or severe according to Accordion severity grading system (Strasberg SM, Linehan DC, Hawkins WG. The Accordion severity grading system of surgical complications. Ann Surg 2009; 250: 177-86.)
Late postoperative complications | Later than 30 days postoperatively
  Late postoperative complications
  Perineal wound healing at 3 months.
  A. Abdominal/donor-site complications
  * superficial wound infection
  * deep wound infection
  * minor wound dehiscence
  * major wound dehiscence
  * abdominal hernia
  * other complications
  B. Perineal complications
  * superficial wound infection
  * deep wound infection
  * minor wound dehiscence
  * major wound dehiscence
  * partial flap loss
  * total flap loss
  * perineal hernia
  * enterocutaneous fistula
  * stricture in neovagina
  * perineal wound dehiscence not related to flap
  * other complications
  C. Other complications
  * incisional hernia
  * parastomal hernia
  * reoperation
  * other complications
  Complications are classified as mild, moderate or severe according to Accordion severity grading system (Strasberg SM, Linehan DC, Hawkins WG. The Accordion severity grading system of surgical complications. Ann Surg 2009; 250: 177-86.)
Quality of life - general | Preoperatively. 3 months and 12 months postoperatively.
  Quality of life - EORTC-QLQ-C30
Quality of life - sexual | Preoperatively. 3 months and 12 months postoperatively.
  Quality of life - EORTC-QLQ-SH22 - excerpt
Abdominal wall strength | Preoperatively. 3 months and 12 months postoperatively.
  Clinical test of abdominal wall strength as described in (Nelson JA et al. Function and strength after free abdominally based breast reconstruction: A 10-year follow- up. Plastic and reconstructive surgery. 2019;143(1):22e-31e.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Frich, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Radiumhospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided